CLINICAL TRIAL: NCT00564005
Title: Mechanisms and Long-term Effects of Separate vs. Coupled Rehabilitation Approaches After Stroke
Brief Title: Mechanism and Efficacy of Rehabilitation Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHRI-EX97-9742PI; 96-0252B
Record Dates: First submitted 2007-11-25; First posted 2007-11-27 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2014-09

CONDITIONS: Cerebrovascular Accidents
Keywords: stroke rehabilitation; cortical reorganization; kinematic analysis
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy; Psychotherapy, Multiple

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): constraint-induced therapy
  Interventions: Other: Constraint-induced therapy (CIT)
- 2 (Experimental): bilateral arm training
  Interventions: Other: Bilateral arm training (BAT)
- 3 (Experimental): combined therapy
  Interventions: Other: Combined therapy (CT)
- Control intervention (Active Comparator)
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Other: Constraint-induced therapy (CIT) — restraint of the unaffected arm and practice of the affected arm
  Arms: 1
Other: Bilateral arm training (BAT) — bilateral symmetric, repetitive arm training
  Arms: 2
Other: Combined therapy (CT) — combined different treatment approaches
  Arms: 3
Behavioral: Control intervention — Conventional treatment program
  Arms: Control intervention

SUMMARY:
Identify the possible mechanisms and the relative effectiveness of existing rehabilitation approaches that target upper extremity deficits of stroke patients on the ground that these approaches are based on neuroplasticity principles and sound motor control theories.

DETAILED DESCRIPTION:
Comparisons of constraint-induced therapy (CIT) vs. bilateral arm training (BIT)vs. combined therapy were made. Stroke patients will receive one of these three approaches and be evaluated pre- and post-treatment. the treatment will last 3 weeks and 5 days per week. The evaluation will include clinical measures of motor function, ADL, and quality of life, kinematic performance, and activation patterns of cortex.

ELIGIBILITY:
Inclusion Criteria:

* a first-ever clinical cerebrovascular accident patients
* at least 6 months post-stroke onset
* premorbid right-hand dominance
* demonstration of Brunnstrom stage III of the affected upper extremity
* no excessive spasticity in the joints of the affected upper extremity

Exclusion Criteria:

* a score of less than 24 on the Mini Mental State Exam
* poor physical conditions that would interfere with participation
* excessive pain in any joint that might limit participation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cortical reorganization and kinematic analysis | 2008-2010

SECONDARY OUTCOMES:
clinical measures at the impairment, activity, participation levels | 2008-2010

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Department of Occupational Therapy, Chang Gung Univ.
Locations (1):
- Chang Gung Memorial Hospital, Kwei-shan, Toayuan County, Taiwan

REFERENCES:
- [Derived] Wu CY, Chen YA, Lin KC, Chao CP, Chen YT. Constraint-induced therapy with trunk restraint for improving functional outcomes and trunk-arm control after stroke: a randomized controlled trial. Phys Ther. 2012 Apr;92(4):483-92. doi: 10.2522/ptj.20110213. Epub 2012 Jan 6. PMID 22228607